CLINICAL TRIAL: NCT01659268
Title: Performance of Nursing Students in the Insertion of Supraglottic Device (Laryngeal Mask): Randomized Controlled Trial on Mannequins.
Brief Title: Performance of Baccalaureate Nursing Students in Insertion of Laryngeal Mask: a Trial in Mannequins
Acronym: LMANURSING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Cesar Eduardo Pedersoli, Performance of baccalaureate nursing students in insertion of supraglottic device (laryngeal mask): a randomized controlled trial in mannequins., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: EERP-2012-LMASIMULATION
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Results first posted 2014-06-02 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2012-12

CONDITIONS: Respiratory Failure
Keywords: teaching; patient simulation; laryngeal masks; baccalaureate nursing education; teaching strategies; simulation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simulation class (Experimental): The students will be submitted a simulation scenario in laboratory with low-fidelity mannequin for 60 minutes, in subgroups of 4-5 students. The simulated condition is a patient in respiratory failure which need of emergency interventions.
  The approach concepts of anatomic, physiology and clinical interventions using LMA will be discussed during simulation.
  Interventions: Other: Simulation class
- Exhibition-dialogued class (Other): Students will be submitted to exhibition-dialogued class with duration of 60 minutes; after this, each subgroup composed of 4-5 students will go to the and practical activity in skill lab using the low-fidelity mannequin for 35 minutes.
  Interventions: Other: Exhibition-dialogued class

INTERVENTIONS:
Other: Simulation class — The students will be submitted a simulation scenario in laboratory with low-fidelity mannequin for 60 minutes, in subgroups of 4-5 students. The simulated condition is a patient in respiratory failure which need of emergency interventions.
  The approach concepts of anatomic, physiology and clinical interventions using LMA will be discussed during simulation.
  Arms: Simulation class
Other: Exhibition-dialogued class — The students randomized to CG will be submitted to exhibition-dialogued class with duration of 60 minutes; after this, will go to practical activity in skill lab using the low-fidelity mannequin with duration of 35 minutes.
  Each subgroup will be composed of 5-6 students for the practice activity which will last 45 minutes.
  Arms: Exhibition-dialogued class

SUMMARY:
The purpose of this study is to compare if there difference in acquisition of knowledge and skills in airway management to baccalaureate nursing students submitted to different learning strategies: exhibition-dialogued class and practical activity in skill lab with low-fidelity mannequin or simulation class with low-fidelity mannequin.

DETAILED DESCRIPTION:
The airway control is priority in patient resuscitation. The Laryngeal Mask Airway (LMA) can minimize complications, establishing a safe airway. Is fundamental to nurse acquired skills to act in emergency situations; the simulation is a important learning tool for this, because allows a realistic environment and allows to student the possibility of training skills.

Hypothesis: There difference in acquisition of knowledge and skills in airway management to baccalaureate nursing students submitted to different learning strategies: classroom lecture-dialogued follow of laboratory activity practice with low-fidelity mannequin or simulation in laboratory with low-fidelity mannequin?

The aim of this study is compare the effect of teaching-learning strategies: classroom lecture-dialogued follow of laboratory activity practice with low-fidelity mannequin or simulation in laboratory with low-fidelity mannequin, in the acquisition of knowledge and skills to baccalaureate nursing. This is a randomized controlled trial, the population is all students of baccalaureate nursing of EERP-USP, eighth period, 69 students in total; the sample will be voluntary and composed for students that accept participate of study. The intervention group (IG) will be submitted to simulation class and the control group (CG)to exhibition-dialogued class, and practical activity in skill lab. The study will have 3 steps:

1. The participants will be recruited with letters and posters, randomized to IG or CG and follow submitted to write pre-test.
2. The GI will submitted to simulation in laboratory and de CG classroom lecture-dialogued follow of laboratory activity practice. The focus will be the airway management with emphasis in LMA.
3. All participants will be submitted to write post test and follow to practice test in simulation scenario, with medium-fidelity mannequin, which simulates human physiologic conditions.

The scenario will have a appraiser with a checklist which performance scores of skills and interventions observed. The activities will be filmed and recorded. To data analysis will be used the SPSS software: descriptive statistics, chi-square test, t-test of Student.

ELIGIBILITY:
Inclusion Criteria:

* student must be in the eighth period of course;
* must be registered regular in the baccalaureate nursing course.

Exclusion Criteria:

* absence in any step of study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cesar E Pedersoli, MSN, Principal Investigator — College of Nursing at Ribeirao Preto - University of Sao Paulo
Locations (1):
- College of Nursing at Ribeirao Preto - University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The strategy of data collect were Workshop "Airway management in emergencies: use of laryngeal mask" which dates of realization 21/11/2012 to 24/11/2012. The disclosure of event were e-mail, site of the institution and posters. Students entries were made through electronic.
Pre-assignment Details: The activities were described for the students in the arrive to the workshop.
Groups:
- Control: The students randomized to CG will be submitted to exhibition-dialogued class with duration of 60 minutes; after this, will go to the and practical activity in skill lab using the low-fidelity mannequin.
  Each subgroup will be composed of 4-5 students for the practice activity which will last 35 minutes.
Period: Overall Study
Arm/Group | Simulation Class | Control
Started | 9 | 8
Completed | 9 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Simulation Class | Control | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (5.2) | 22.6 (1.69) | 24.4 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Brazil | 9 | 8 | 17

OUTCOME MEASURES:

1. Primary Outcome: Scores in Pre and Post-test, Number of Participants Successfully Completing the Overall Performance Simulated Scenario(OSCE).
Description: Score obtained in pre and post-test written, time to obtain the first effective ventilation (chest expansion through adequate ventilation on the mannequin), number of attempts to insert the LMA in the simulation scenario (OSCE).
  Pre-test: 20 questions with score of 0.5 points each - minimum score=0 points and maximum score=10 points. Score 5-7 points was considered satisfactory; scores between 7-8 points was considered good performance; above 8 points excellent.
  Post-test: 20 questions with score of 0.5 points each - minimum score=0 points and maximum score=10 points. Score 5-7 points was considered satisfactory; scores between 7-8 points was considered good performance; above 8 points excellent.
  OSCE: instrument with total of 10 skills - each skill was subdivided in 4-5 activities (0.2-0.25 points each) - poor performance was score < 5.0; satisfactory performance 5.0-7.0; good 7.0-8.5 and excellent above 8.5 points.
Time Frame: Pretest: 40 minutes; Post-test: 40 minutes; OSCE: 10 minutes
Population: The number of participants result of students that signed up in the workshop.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Simulation Class | Control
Number analyzed (Participants) | 9 | 8
units on a scale
  Pre-test | 6.6 (1.0) | 6.5 (0.5)
  Postest | 8.6 (1.1) | 8.4 (0.8)
  OSCE's score | 8.4 (0.89) | 7.8 (0.52)

2. Secondary Outcome: Time for Acquisition of First Effective Ventilation, Adequate Tidal Volume and Stabilization of Patient.
Description: Time of achievement to first effective ventilation and tidal volume (adequate chest expansion).
  Stabilization of mannequin parameters (spO2 e HR).
Time Frame: 10 minutes (600 sec)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Simulation Class | Control
Number analyzed (Participants) | 9 | 8
seconds | 428.1 (143.6) | 426.5 (172)

3. Secondary Outcome: Number of Attempts to Insertion of LMA
Description: Number of attempts for insertion of LMA and obtainment of effective ventilation.
Time Frame: 10 minutes (total time of scenario)
Measure: Mean (Standard Deviation); unit: attempts
Arm/Group | Simulation Class | Control
Number analyzed (Participants) | 9 | 8
attempts | 1.56 (0.63) | 1.63 (0.74)

4. Primary Outcome: Time to Conclusion of Simulation Scenario (OSCE)
Description: This result present the total time for execution of simulation scenario (OSCE) by the students.
Time Frame: 10 minutes
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Simulation Class | Control
Number analyzed (Participants) | 9 | 8
seconds | 520.3 (157) | 479.8 (183.3)

ADVERSE EVENTS:
Arm/Group | Simulation Class | Control
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8
Other Adverse Events (participants affected / at risk) | 0/9 | 0/8

LIMITATIONS AND CAVEATS:
The limitations of this study are due to the small number of participants in the sample, even after running wide dissemination workshop for print and electronic media with students nursing institution involved in research.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No